CLINICAL TRIAL: NCT02968667
Title: The Effectiveness of Hopelessness and Helplessness on Recovery Rate Among People Diagnosed With Schizophrenia
Brief Title: The Impact of a Helplessness and Recovery of an Empowerment Intervention on People Diagnosed With Schizophrenia: Findings From a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fakeeh College for Medical Sciences (Other)
Responsible Party: Principal Investigator, Abd Alhadi Hasan, Assistant professor, Fakeeh College for Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FakeehCMS
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention group received 6 weeks of empowerment program
  Interventions: Behavioral: Empowerment
- Treatment as usual (No Intervention): Medications

INTERVENTIONS:
Behavioral: Empowerment — 6 weeks of empowerment program and supported face to face discussion
  Arms: Intervention

SUMMARY:
A randomized controlled trial was conducted from November 2015 and May 2016 with 112 participants of people diagnosed with schizophrenia. Participants aged 18 years or older with Diagnostic Statistical Manual (DSM-V) schizophrenia or schizoaffective disorder from outpatient mental health clinics in Jordan, were randomly assigned participants either to receive 6 weeks of a booklet form of intervention with face to face discussion, and treatment as usual (TAU) (intervention, n = 56), or TAU (control, n = 56). Participants were assessed at baseline, immediately post-intervention (post-treatment1) and at three months follow-up. The primary outcome measure was change in helplessness score . Secondary outcomes for PDwS were psychiatric symptoms, recovery rate and quality of life.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted from November 2015 and May 2016 with 112 participants of people diagnosed with schizophrenia. Participants aged 18 years or older with DSM-V schizophrenia or schizoaffective disorder from outpatient mental health clinics in Jordan, were randomly assigned participants either to receive 6 weeks of a booklet form of intervention with face to face discussion, and treatment as usual [TAU] (intervention, n = 56), or TAU (control, n = 56). Participants were assessed at baseline, immediately post-intervention (post-treatment1) and at three months follow-up. The primary outcome measure was change in helplessness score . Secondary outcomes for PDwS were psychiatric symptoms, recovery rate and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 16 years or more
* Able to read and write in an Arabic
* Able to consent
* Diagnosed with schizophrenia
* Volunteers

Exclusion Criteria:

* Learning disability
* Not able to read or write

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Modified Learned Helplessness | Up to 6 months
  Outcome was measured at baseline (November) and immediately post intervention (February) and at three months follow up (May)

SECONDARY OUTCOMES:
Psychiatric symptoms | Up to 6 months
  Outcome was measured at baseline (November) and immediately post intervention (February) and at three months follow up (May)
recovery assessment scale | Up to 6 months
  Outcome was measured at baseline (November) and immediately post intervention (February) and at three months follow up (May)
Empowerment level | Up to 6 months
  Outcome was measured at baseline (November) and immediately post intervention (February) and at three months follow up (May)
Quality of life | Up to 6 months
  Outcome was measured at baseline (November) and immediately post intervention (February) and at three months follow up (May)